CLINICAL TRIAL: NCT01591044
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of Two Doses of Inhaled R940343 in Patients With Mild to Moderate Allergic Asthma
Brief Title: A Safety and Efficacy Study of Inhaled R940343 in Patients With Mild to Moderate Asthma
Acronym: SITAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-940343-004
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- R940343 2mg, 2 puffs bid (Active Comparator): R343 2mg, 2 puffs bid
  Interventions: Drug: R940343 2mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- R940343 1mg, 1 puff bid (Active Comparator): R343 1mg, 1 puff bid
  Interventions: Drug: R940343 1mg

INTERVENTIONS:
Drug: Placebo — 1 puff bid or 2 puffs bid
  Arms: Placebo
Drug: R940343 1mg — R343 1mg, 1 puff bid
  Other Names: R343
  Arms: R940343 1mg, 1 puff bid
Drug: R940343 2mg — R343 2mg, 2 puffs bid
  Other Names: R343
  Arms: R940343 2mg, 2 puffs bid

SUMMARY:
The purpose of this study is to determine the safety, efficacy and tolerability of R940343 in the treatment of mild to moderate asthma.

DETAILED DESCRIPTION:
The study is a multi-center, randomized, double-blind, placebo-controlled, parallel group study comparing 2 doses of inhaled R343 bid to placebo over 8 weeks in patients with mild to moderate allergic asthma. Patients who meet specific inclusion and exclusion criteria after an initial screening evaluation and a single-blind, run-in period will be randomized to receive either R343 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of asthma
* Ability to perform spirometry

Exclusion Criteria:

* Chronic obstructive pulmonary disease or bronchiectasis
* Upper or lower respiratory infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Grossbard, MD, Study Director — Rigel Pharmaceuticals,Inc.
Locations (59):
- United States (51):
  - California Research Medical Group, Inc, Fullerton, California
  - Allergy Medical Clinic Research Division, Los Angeles, California
  - California Allergy & Asthma Medical Group, INC, Los Angeles, California
  - Southern California Institute for Respiratory Diseases, Inc., Los Angeles, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - CHOC PSF, AMC, Division of Allergy, Asthma & Immunology, Orange, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy Associates Medical Group. Inc., San Diego, California
  - Allergy & Asthma Med Group/Research Center, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley, San Jose, California
  - Bensch Research Associates, Stockton, California
  - Colorado Allergy and Asthma Clinic, PC, Centennial, Colorado
  - Asthma & Allergy Associates, PC, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - Colorado Allergy & Asthma Centers, PC, Denver, Colorado
  - Florida Center for Allergy & Asthma Research, Aventura, Florida
  - Accelovance, Melbourne, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Georgia Pollens Clinical Research Centers, Inc., Albany, Georgia
  - Idaho Allergy DBA Idaho Research, Eagle, Idaho
  - Sneeze, Wheeze & Itch Associates, Normal, Illinois
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Respiratory Medicine Researh Institute of Michigan, Ypsilanti, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Inc., Plymouth, Minnesota
  - Clinical Research of The Ozarks, Inc., Columbia, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Clinical Research Group of Montana PLLC, Bozeman, Montana
  - The Asthma & Allergy Center, Bellevue, Nebraska
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Allergy Consultants, PA, Verona, New Jersey
  - New York Pulmonary Associates, P.C., New York, New York
  - Allergy Asthma Immunology of Rochester (AAIR), Rochester, New York
  - Peters Medical Research, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy & Asthma Research Group, Eugene, Oregon
  - Clinical Research Inst. of Southern Oregon, PC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy, Asthma and Uticaria Center of Charleston, Charleston, South Carolina
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Western Sky Medical Research, Inc., El Paso, Texas
  - Live Oak Allergy & Asthma Clinic, Live Oak, Texas
  - Allergy & Asthma Care of Waco, PA, Waco, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - ASTHMA, Inc., Seattle, Washington
  - MultiCare Pulmonary Specialists, Tacoma, Washington
- Canada (8):
  - Joseph Greenbaum, MD, Hamilton, Ontario
  - Cheema Research, Inc., Missassauga, Ontario
  - Niagara Clinical Research, Niagara Falls, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Pulmonary Care Clinic, Toronto, Ontario
  - Primary Care Lung Clinic, Toronto, Ontario
  - Dynamik Research, Inc., Pointe-Claire, Quebec
  - Centre De recherche Appliquee en Allergie DeQuebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- R940343 2mg, 2 Puffs Bid: R343 2mg, 2 puffs bid
  R940343: R343 1mg, 1 puff bid R343 2mg, 2 puffs bid
- R940343 1mg, 1 Puff Bid: R343 1mg, 1 puff bid
  R940343: R343 1mg, 1 puff bid R343 2mg, 2 puffs bid
Period: Overall Study
Arm/Group | R940343 2mg, 2 Puffs Bid | Placebo | R940343 1mg, 1 Puff Bid
Started | 101 | 100 | 100
Completed | 94 | 91 | 96
Not Completed | 7 | 9 | 4

BASELINE CHARACTERISTICS:
Population: For the purpose of analysis, participants randomized to the two different dosage levels of the placebo were considered a single Arm/Group.
Groups:
- Placebo: Placebo: 1, 1 puff bid or 2, 2 puffs bid
- Total: Total of all reporting groups
Arm/Group | R940343 2mg, 2 Puffs Bid | Placebo | R940343 1mg, 1 Puff Bid | Total
Number analyzed (Participants) | 101 | 100 | 100 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.5) | 38.3 (12.6) | 39.3 (12.8) | 39.1 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 58 | 55 | 164
  Male | 50 | 42 | 45 | 137

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1
Description: Change from baseline in pre-BD FEV1 (% predicted) at Week 8.
Time Frame: Baseline and Week 8
Population: All efficacy endpoints were analyzed based on the intent to treat population consisting of all randomized patients.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | R940343 2mg, 2 Puffs Bid | Placebo | R940343 1mg, 1 Puff Bid
Number analyzed (Participants) | 101 | 100 | 100
percentage of change | -0.40 (8.56) | 0.69 (9.31) | -0.59 (8.75)

ADVERSE EVENTS:
Time Frame: The adverse event reporting period begins with the first dose of study drug and ends with the final study follow-up visit (week 9).
Arm/Group | R940343 2mg, 2 Puffs Bid | Placebo | R940343 1mg, 1 Puff Bid
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 36/101 | 48/100 | 26/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R940343 2mg, 2 Puffs Bid (N=101) | Placebo (N=100) | R940343 1mg, 1 Puff Bid (N=100)
Eye Disorders (Eye disorders) | 1 (1) | 1 (1) | 1 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ear and Labyrinth Disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
General Disorders and Administration Site Conditions (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 20 (20) | 26 (26) | 9 (9)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Investigations (Investigations) | 3 (3) | 3 (3) | 1 (1)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9) | 8 (8)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less